CLINICAL TRIAL: NCT04620551
Title: Adaptive Neurostimulation to Restore Sleep in Parkinson's Disease: An Investigation of STN LFP Biomarkers in Sleep Dysregulation and Repair
Brief Title: Adaptive Neurostimulation to Restore Sleep in Parkinson's Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Stanford University (Other); University of Pennsylvania (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0120-20-FB
Record Dates: First submitted 2020-11-02; First posted 2020-11-09 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease; Sleep Fragmentation
MeSH Terms: conditions — Parkinson Disease; Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- PD with DBS (Experimental): Patients with Parkinson's Disease who opt for DBS surgery and consent to participate in the sleep study.
  Interventions: Device: Sub-clinical stimulation

INTERVENTIONS:
Device: Sub-clinical stimulation — The third night of recording will involve sub-clinical thresholds of stimulation in all subjects.

SUMMARY:
Parkinson's disease (PD) is a neurodegenerative disorder that leads to both motor and non-motor symptoms. Therapies have been developed that effectively target the motor symptoms. Non-motor symptoms are far more disabling for patients, precede the onset of motor symptoms by a decade, are more insidious in onset, have been less apparent to clinicians, and are less effectively treated. Sleep dysfunction is oftentimes the most burdensome of the non-motor symptoms. There are limited options for treating sleep dysfunction in PD, and the mainstay of therapy is the use of sedative-hypnotic drugs without addressing the underlying mechanisms. Patients with PD who demonstrate significant motor fluctuations and dyskinesia are considered for subthalamic nucleus (STN) deep brain stimulation (DBS) surgery. Several studies have reported that STN-DBS also provides benefit for sleep dysregulation. Additionally, local field potentials recorded from STN DBS electrodes implanted for the treatment of PD, have led to the identification of unique patterns in STN oscillatory activity that correlate with distinct sleep cycles, offering insight into sleep dysregulation. This proposal will leverage novel investigational DBS battery technology (RC+S Summit System; Medtronic) that allows the exploration of sleep biomarkers and prototyping of closed-loop stimulation algorithms, to test the hypothesis that STN contributes to the regulation and disruption of human sleep behavior and can be manipulated for therapeutic advantage. Specifically, in PD patients undergoing STN-DBS, the investigators will determine whether STN oscillations correlate with sleep stage transitions, then construct and evaluate sensing and adaptive stimulation paradigms that allow ongoing sleep-stage identification, and induce through adaptive stimulation an increase in duration of sleep stages associated with restorative sleep.

DETAILED DESCRIPTION:
Although STN-DBS is routinely used to treat PD motor symptoms, several studies have reported that STN-DBS also provides benefit for sleep dysregulation through normalization of sleep architecture. In our previous work, using local field potentials (LFP) recorded from STN DBS electrodes implanted for the treatment of PD, unique spectral patterns in STN oscillatory activity were identified that correlated with distinct sleep cycles, offering insight into sleep dysregulation. These findings were used to construct an Artificial Neural Network (ANN) that can accurately predict sleep stage. Building on this work with the use of new DBS battery technology that allows exploration of potential biomarkers and prototyping of closed-loop algorithms, the investigators will test the hypothesis that STN-a highly interconnected node within the basal ganglia- contributes to the regulation and disruption of human sleep behavior and can be manipulated for therapeutic advantage.

This is the first part, Aim 1, of a two-part study. Investigators will enroll 20 subjects for Aim 1 of this study and 20 subjects for Aim 2, with 10 subjects enrolled at each clinical site for each aim (University of Nebraska Medical Center and Stanford University Medical Campus). In Aim 1, subjects will undergo standard-of-care STN DBS lead implantation surgery for the treatment of PD. They will return 3 weeks later to the in-patient Sleep Lab for 3 nights of STN LFP recordings with concurrent PSG, EMG, EOG, actigraphy, and video-EEG. The first two nights of recording will be used to establish a physiological sleep baseline for each patient. The third night of recording will involve sub-clinical thresholds of stimulation in all subjects, in an effort to favorably alter sleep-stage duration, so that NREM and REM-3 are prolonged. As a secondary outcome, subjects will be asked to complete a sleep questionnaire for all three nights, sleep during which stimulation occurred will be compared to the preceding two nights. Data collected during all three nights of recordings will be used to predict sleep stage identity from the LFPs recorded within STN, with the ground truth for each sleep stage provided by sleep-expert evaluated PSG. These data will also be used to identify the optimal sub-clinical threshold current amplitude and sleep-stage timing for adaptive stimulation to improve sleep. The stimulation algorithm developed in Aim 1 will be implemented in the second part of the study, Aim 2, to provide adaptive stimulation to subjects during nighttime sleep, over the course of 3 weeks of in-home sleep.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent for this study
* Diagnosis of Idiopathic Parkinson's disease with motor symptoms that have been present for a minimum of 4 years
* Motor symptoms are severe enough, despite optimized medical therapy, to warrant surgical implantation of DBS
* UPDRS-III score off medication between 20 and 80, and an improvement in UPDRS-III score on medications of at least 30%, or patients with tremor-dominant PD (score >/= 2 on UPDRS-III tremor sub-score)-or tremor in addition to other motor symptoms-that is treatment-resistant and results in significant functional disability
* Appropriate trials of oral PD medications have resulted in inadequate relief of motor symptoms
* Absence of abnormalities on brain MRI suggestive of an alternate diagnosis or serving as a contraindication to surgery
* Absence of significant cognitive deficits or significant depression (BDI-II score > 20) on formal Neuropsychological Testing
* Age 21 - 80 years

Exclusion Criteria:

* Coagulopathy, uncontrolled hypertension, history of seizures, heart disease, inability to undergo general anesthesia
* Pregnancy
* Significant untreated depression (BDI-II score > 20)
* Personality or mood disorder symptoms that Study Personnel believe will interfere with study requirements
* Patients requiring ongoing treatment with ECT, rTMS, or diathermy
* Pre-existing implanted stimulation system (e.g., cochlear implant, cardiac pacemaker, defibrillator, neuro-stimulator for indication other than Parkinson's disease) or ferromagnetic metallic implant
* Prior intracranial surgery
* History of, or active, drug or alcohol abuse
* Meets criteria for PD with Mild Cognitive Impairment (PD-MCI), as defined by Performance > 2 standard deviations below appropriate norms on tests from 2 or more of the following cognitive domains: Attention, Executive Function, Language, Memory, and Visuospatial Ability
* Patients with Restless Leg Syndrome

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Sleep stage duration and transitions | Years 1-2
  We will measure pre- vs. post-stimulation impact on (1) LFP spectral composition; (2) sleep episode-specific change in duration; and (3) stimulation-induced latency to transition to next sleep episode.

SECONDARY OUTCOMES:
Sleep Quality | Years 1-2
  Study participants will complete the Pittsburgh Sleep Diary as a measure of self-reported sleep quality and sleep disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Aviva Abosch, MD, PhD, Study Director — University of Nebraska; Casey Halpern, MD, Principal Investigator — Stanford University; Clete Kushida, MD, PhD, Principal Investigator — Stanford University; John Thompson, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Das R, Gliske SV, West LC, Summers MO, Tang S, Hirt L, Maroni D, Halpern CH, Thompson JA, Kushida CA, Abosch A. Sleep macro-architecture in patients with Parkinson's disease does not change during the first night of neurostimulation in a pilot study. J Clin Sleep Med. 2024 Sep 1;20(9):1489-1496. doi: 10.5664/jcsm.11180. PMID 38652493
- [Derived] West LC, Summers M, Tang S, Hirt L, Halpern CH, Maroni D, Das R, Gliske SV, Abosch A, Kushida CA, Thompson JA. Evaluation of consensus sleep stage scoring of dysregulated sleep in Parkinson's disease. Sleep Med. 2023 Jul;107:236-242. doi: 10.1016/j.sleep.2023.04.031. Epub 2023 May 18. PMID 37257366